CLINICAL TRIAL: NCT02132546
Title: Spectrophotometric Evaluation of Chlorhexidine Pigmentations After Periodontal Flap Surgery: a Prospective Randomized Clinical Trial
Brief Title: Spectrophotometric Evaluation of Chlorhexidine Pigmentations After Oral Surgery: a Prospective Randomized Clinical Trial
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: dott. Lorenzo Bevilacqua (Other)
Responsible Party: Sponsor-Investigator, dott. Lorenzo Bevilacqua, DDS, MS, University of Trieste
Organization: University of Trieste (Other)
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: AAA-0001-TS
Record Dates: First submitted 2014-04-30; First posted 2014-05-07 (Estimated); Last update posted 2014-05-07 (Estimated); Status verified 2014-04

CONDITIONS: Staining Effect of Chlorhexidine
MeSH Terms: interventions — Chlorhexidine

STUDY DESIGN:
Who Masked: Participant, Care Provider

ARMS (3):
- Chlorhexidine 0,2% (Experimental): After surgery, the patient was given instruction following the post-operative protocol. Oral hygiene with toothbrush and dental floss was suspended only in the area that underwent periodontal surgery and the patient was given an anonymous bottle of mouthwash. According to random assignment (random generator, www.random.org), the bottle contained 0.2% CHX.
  Interventions: Drug: Chlorhexidine
- Chlorhexidine 0,2% with ADS (Experimental): After surgery, the patient was given instruction following the post-operative protocol. Oral hygiene with toothbrush and dental floss was suspended only in the area that underwent periodontal surgery and the patient was given an anonymous bottle of mouthwash. According to random assignment (random generator, www.random.org), the bottle contained 0.2% CHX with ADS.
  Interventions: Drug: Chlorhexidine
- Chlorhexidine 0,12% (Experimental): After surgery, the patient was given instruction following the post-operative protocol. Oral hygiene with toothbrush and dental floss was suspended only in the area that underwent periodontal surgery and the patient was given an anonymous bottle of mouthwash. According to random assignment (random generator, www.random.org), the bottle contained 0.12% CHX.
  Interventions: Drug: Chlorhexidine

INTERVENTIONS:
Drug: Chlorhexidine

SUMMARY:
The aim of this clinical trial was to evaluate through a clinical spectrophotometric analysis the staining side effect of a 0.2% CHX mouthwash containing an anti discoloration system (ADS) compared with a 0.12% and a 0.2% CHX alone mouthwash after periodontal surgery. The efficacy of the products and the patient's opinion and acceptance were also assessed.

ELIGIBILITY:
Inclusion Criteria:

* Good general health conditions without a medical history of medication that might interfere with periodontal tissues
* Good plaque control (FMPS ≤ 25%) and low levels of infection (FMBS ≤ 25%)
* Need for periodontal surgery

Exclusion Criteria:

* Smokers
* Allergy to CHX
* Lack of written informed consent

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2011-02; Primary Completion 2011-10 (Actual); Study Completion 2012-09 (Actual)

PRIMARY OUTCOMES:
Change in ΔE before and after the use of chlorhexidine | Change from Baseline of ΔE after the use of chlorhexidine mouthrinses; change from Baseline of ΔE after the use of chlorhexidine mouthrinses at 1 week; change from Baseline of ΔE after the use of chlorhexidine mouthrinses at 2 weeks
  Change in ΔE before and after the use of chlorhexidine (ΔE is a measurement used to indicate how much a color deviates from an accepted standard. Perfect color has a ΔE of zero.)

CONTACTS AND LOCATIONS:
Locations (1):
- Ospedale Maggiore, Trieste, Italy, Italy